CLINICAL TRIAL: NCT04065360
Title: Effectiveness of Group Cognitive Behavioural Family Intervention (CBFI) for People With Schizophrenia and Their Families: A Mixed-method Study
Brief Title: Group Cognitive Behavioural Family Intervention (CBFI) for People With Schizophrenia and Their Families
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chak Fai Ma, Registered Nurse (Psychiatric), Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBFI
Record Dates: First submitted 2019-08-17; First posted 2019-08-22 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Psychosis
Keywords: Schizophrenia; Psychosis; Family intervention; Cognitive behavioural therapy; CBT
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural family intervention (Experimental)
  Interventions: Behavioral: Group Cognitive behavioural family intervention (CBFI)
- Usual group psychoeducation (Active Comparator)
  Interventions: Behavioral: Usual group psychoeducation

INTERVENTIONS:
Behavioral: Group Cognitive behavioural family intervention (CBFI) — four-week, four-session CBT-based family intervention programme
  Arms: Cognitive behavioural family intervention
Behavioral: Usual group psychoeducation — Treatment as usual in the institution studied
  Arms: Usual group psychoeducation

SUMMARY:
Cognitive behavioural family intervention (CBFI) is a brief psychosocial intervention that incorporates the model of cognitive behavioural therapy (CBT) into the family context. It builds upon the current trend of family interventions/psychoeducation with refocusing on the cognitive model within the family interpersonal relationship. Existing literature indicates that CBFI may be effective in improving positive and negative symptoms of people diagnosed with schizophrenia immediately following the programme. This mixed-method is to evaluate the feasibility and effectiveness of a CBFI programme for people with schizophrenia and their families in a local context. The findings may accumulate more evidence that CBFI is a brief and effective psychosocial intervention that is adapted to Hong Kong clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Service users

* Diagnosis of schizophrenia-spectrum disorders, based on clinical judgement by the treating clinicians
* Aged 18-65
* Able to communicate in Cantonese

Family caregivers

* Aged above 18
* Living with service users
* Able to communicate in Cantonese
* Nominated by the service users

Exclusion Criteria:

Service users

* Having co-morbidity of learning disability
* Organic/neurological conditions
* Substance misuse disorder

Family caregivers

* Having active psychiatric conditions
* Looking after more than one family member suffering from chronic physical or mental illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative feedback from the clinicians of the concerned wards | Immediate posttreatment
  Programme evaluation interview

SECONDARY OUTCOMES:
Positive symptoms of service users | Immediate posttreatment
  Psychotic Symptoms Rating Scales (PSYRATS); 11-item hallucination subscale ranging from 0 to 44; 6-item delusion subscale ranging from 0 to 24
Negative symptoms of service users | Immediate posttreatment
  Brief Negative Symptom Scale (BNSS); 13-item ranging from 0 to 78
Expressed emotion by service users | Immediate posttreatment
  Concise Chinese Level of Expressed Emotion Scale (CCLEES); 12-item ranging from 12 to 48
Caregiving experience by family caregivers | Immediate posttreatment
  Chinese version of Experience of Caregiving Inventory (CECI); 66-item ranging from 0 to 264
Perceived care burden by family caregivers | Immediate posttreatment
  Family Burden Interview Schedule (FBIS); 25-item ranging from 0 to 50
Mood disturbance by family caregivers | Immediate posttreatment
  Hospital Anxiety and Depression Scale (HADS); 7-item depression subscale ranging from 0 to 21; 7-item anxiety subscale ranging from 0 to 21
Qualitative feedback from the service users and their families | Immediate posttreatment
  Semi-structured focus group interview

CONTACTS AND LOCATIONS:
Overall Officials: Chak Fai Ma, MSc, Principal Investigator — Kwai Chung Hospital
Locations (1):
- Kwai Chung Hospital, Hong Kong, Hong Kong